CLINICAL TRIAL: NCT03797508
Title: Biochemical Versus Ultrasound Findings as Predictors of Fetal Loss in Cases of First Trimester Threatened Miscarriage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, amany abdel monem mahmoud, Egypt Cairo, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: us laboratory miscarriage
Record Dates: First submitted 2019-01-06; First posted 2019-01-09 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Abortion Threatened
MeSH Terms: conditions — Abortion, Threatened | interventions — Ultrasonography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- threatened miscarriage (Other): ultrasound ,CA125,progesterone
  Interventions: Diagnostic Test: ultrasound

INTERVENTIONS:
Diagnostic Test: ultrasound — To evaluate the accuracy of ultrasound findings in comparison to serum CA125and progesterone in predicting fetal demise in cases of first trimester threatened miscarriage.
  Other Names: progesterone; CA125

SUMMARY:
Threatened miscarriage occurs in about one-fifth of pregnancies with an estimated miscarriage rate of 3-16% after successful demonstration of fetal cardiac activity. Various biochemical markers have been studied previously to predict the outcome of threatened miscarriage; However, the results have been conflicting. Several studies have documented that a slow embryonic heart rate at 6.0-7.0 Weeks' gestation is associated with a high rate of first trimester fetal demise.

our aim: To evaluate the accuracy of ultrasound findings in comparison to serum CA125 and progesterone in predicting fetal demise in cases of first trimester threatened miscarriage.

Will this pregnancy be continued after the first trimester or not?

DETAILED DESCRIPTION:
we are comparing between the accuracy of vaginal ultra sound versus serum progesterone level and serum CA 125 level in predicting of fetal demise in cases of threatened miscarriage three vaginal ultrasounds will be done ) the first one will be done at six to eight weeks of pregnancy to the patients who fulfill the criteria in this us we will make sure that the cardiac pulsations are present and measure the following:

1. the fetal heart rate,
2. the crown rump length
3. gestational sac diameter
4. yolk sac diameter. b) The second ultra sound will be after two weeks from the first one to follow up the patient for pregnancy survival, take the same measures again and correlate them with the results of laboratory investigations to select the investigation which is most accurate in anticipating outcome in cases of threatened abortion.

C) the third one will be at the end of first trimester (13 weeks) to ensure fetal viability.

. embryonic bradycardia and absence of yolk sac or smaller yolk sac than expected for any given gestational age are prognostic factors of poor pregnancy outcome in the first 12 weeks of pregnancy women with small for age gestational sac are more prone to have miscarriage we will do laboratory investigation in the form of A) Serum progesterone: low maternal P levels have been useful in predicting spontaneous abortion in threatened pregnancies with a sensitivity of 80% (<10 ng /mL) so, this will be our cutoff value. B) Serum CA 125 :we will take a level of 51.5 as cut off value.this is the upper level of normal we will do them once when the patient presents to us.

ELIGIBILITY:
Inclusion Criteria:

* Singleton Pregnancy.
* Age20-35years.
* Gestational age between6 to 8weeks.
* Threatened miscarriage is diagnosed by vaginal bleeding, closed cervix and positive fetal life.
* Patients who are sure of their dates (three regular menstrual cycles before conception without the use of hormonal contraception.

Exclusion Criteria:

Patients with recurrent miscarriage or pregnancy of unknown location (PUL).

* Patients had ovulation induction medications or on progesterone treatment.
* Patients with past medical history of diabetes mellitus or chronic hypertension.
* Patients who are unsure of the last menstrual period date or with irregular menstrual cycle.
* Pregnancy associated with presence of ovarian cyst.
* Molar pregnancy.
* Those who had a history of maternal disease which would cause an increase in CA-125level. These diseases include chronic pelvic infection, endometriosis, myoma uteri, endometrioma and lung, kidney and hepatic diseases.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
ultra sound | the 12th week of gestation
  presence of fetal heart rate

CONTACTS AND LOCATIONS:
Overall Officials: amany a mahmoud, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt